CLINICAL TRIAL: NCT03523650
Title: Oral Propanolol for Surgically Inaccessible Cerebral and Spinal Cavernous Malformations
Brief Title: Oral Propanolol for Surgically Inaccessible Cavernous Malformations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Yashar Kalani, MD, Co-Director of Neurovascular Surgery, Director of Skull Base Surgy and Director of Stroke Center, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20195
Record Dates: First submitted 2018-04-13; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Cavernous Malformations,Cerebral and/or Spinal
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Propranolol Group (Experimental): Group 1: Propranolol - group of randomized patients will receive one propranolol pill tid for 36 months.
  Interventions: Drug: Propranolol Oral Tablet
- Group 2: Placebo Group (Placebo Comparator): Group 2: Placebo - group of randomized patients will receive one placebo pill tid for 36 months.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Propranolol Oral Tablet — A randomized group of patients with cerebral or spinal cavernous malformations, will receive a Propranolol Oral tablets, tid, for 36 months.
  Arms: Group 1: Propranolol Group
Drug: Placebo Oral Tablet — A randomized group of patients with cerebral or spinal cavernous malformations, will receive a Placebo Oral Tablet, tid, for 36 months.
  Arms: Group 2: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the role of propranolol as an alternative treatment for cavernous malformation in patients that may not be ideal candidates for surgery.

DETAILED DESCRIPTION:
Patients between the ages of 1 and 80 years of age, that have been diagnosed with a spinal or cerebral cavernous malformation(s) that can not be surgically treated, will be enrolled in this randomized study. All eligible patients will be enrolled in one of two groups. Group 1 will receive oral propranolol tablets 3 times a day for 36 months. Group 2 will receive oral placebo tablets 3 times per day for 36 months. Prior to beginning treatment, all imaging, including MRIs, will be evaluated. During the first visit a blood sample will be collected for genomic analysis. Patients will return to clinic every 6 months. Each time the patient returns to clinic monitoring of how the patient is feeling and evaluation of how the patient is tolerating the propranolol will take place. At the end of the three years, evaluators will determine if the propranolol was able to stop the growth of the cavernous malformation and change the imaging features of the lesion on MRI. Once the study is completed patients will no longer receive the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of isolated or familial cavernous malformation syndrome:

   * symptomatic cavernous malformation not amenable to surgical resection.
   * familial cavernous malformation with seizure, other neurological symptom or surgically inaccessible lesion.
2. Written and informed consent obtained prior to study enrollment.
3. Subject is able and willing to return for outpatient visits.
4. Negative pregnancy test at time of enrollment for women and child-bearing potential.

Exclusion Criteria:

1. Age less than 1 year-old.
2. Propranolol allergy or allergy to other b-blockers.
3. Estimated life expectancy of less than 1 year.
4. History of severe anemia, cardiac dysfunction, or diabetes.
5. A psychiatric or substance abuse problem that may interfere with study compliance.
6. Pregnant and lactating women.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Number of symptomatic and silent hemorrhages on MRI | 36 months
  Using MRI imaging the size of the cavernous malformation will be measured. The primary outcome is the number of symptomatic and silent hemorrhages as assessed by review of a fine-cut, axial T2-weighted MRI obtained at each visit.

SECONDARY OUTCOMES:
Rate of de novo lesion formation; changes in rate of breakthrough seizures or other neurological deficits | 36 months
  The secondary outcome is the rate of de novo lesion formation; changes in rate of breakthrough seizures or other neurological deficits; quality of life measured using the SF-36 at each visit, patient satisfaction with treatment; and the incidence of treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Yashar Kalani, MD, PHD, Principal Investigator — University of Virginia Medical Center
Locations (1):
- Univeristy of Virginia, Charlottesville, Virginia, United States